CLINICAL TRIAL: NCT05080348
Title: Effectiveness of Preoperative iPACK on Postoperative Pain From Hamstring Autograft for ACL Repair
Brief Title: Effectiveness of iPACK on Postoperative Pain From Hamstring Autograft Following ACL Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brenton Alexander (Other)
Responsible Party: Sponsor-Investigator, Brenton Alexander, Associate Physician, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: iPACK ACL Hamstring Autograft
Record Dates: First submitted 2021-09-07; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Pain, Postoperative; ACL Injury; Anesthesia, Local; Opioid Use
MeSH Terms: conditions — Pain, Postoperative; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Randomized double blind placebo controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patient will not know which group they are in as they will be injected with either SHAM or Intervention group, which the pharmacy will create. As a result, the anesthesiologist performing the injection and the intraoperative anesthesiologist will also not know if the patient received a SHAM or intervention injection. This will also apply to the PACU nurse. The person performing the data analysis will know which patients received the intervention, as this is required for data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine iPACK (Active Comparator): Patient will receive standard of care for perioperative pain management. In addition, they will receive a single preoperative injection of 20cc of 0.25% Ropivacaine with 1:400,000 epinephrine in the Interspace between the Popliteal Artery and Capsule of the Knee (iPACK).
  Interventions: Procedure: Ropivacaine iPACK Injection
- Normal Saline iPACK (Sham Comparator): Patient will receive standard of care for perioperative pain management. In addition, they will receive a single preoperative injection of 20cc of 0.9% Normal Saline in the Interspace between the Popliteal Artery and Capsule of the Knee (iPACK).
  Interventions: Procedure: Normal Saline iPACK Injection

INTERVENTIONS:
Procedure: Ropivacaine iPACK Injection — Injection of 20mL of 0.25% Ropivacaine with 1:400,000 Epinephrine between in the Interspace between the Popliteal Artery and the Capsule of the Knee (iPACK) using ultrasound guidance at the level of the femoral condyles
  Arms: Ropivacaine iPACK
Procedure: Normal Saline iPACK Injection — Injection of 20mL of 0.9% Normal Saline between in the Interspace between the Popliteal Artery and the Capsule of the Knee (iPACK) using ultrasound guidance at the level of the femoral condyles
  Arms: Normal Saline iPACK

SUMMARY:
Patients undergoing ACL repair with hamstring autograft frequently develop significant post operative pain at the hamstring grafting site. This pain is within the distribution of a commonly used regional nerve block, the Interspace between the popliteal artery and capsule of the knee (iPACK). The investigators plan to randomize consenting patients to either receiving a SHAM injection of normal saline or to an interventional group of long acting local anesthetic (Ropivacaine) injected in the popliteal fossa between the popliteal artery and capsule of the knee (iPACK). Both groups of patients will receive standard of care with respect to perioperative pain management, which includes a preoperative adductor canal nerve block and preoperative acetaminophen administration. Dual primary endpoints of postoperative pain scores and mean postoperative opioid use will be retrieved and compared between groups. Additional secondary endpoints will be PACU length of stay, PACU opioid use, POD1 opioids use, and POD1 pain scores (best, worst, average).

ELIGIBILITY:
Inclusion Criteria:

* Undergoing ACL surgery with expected Hamstring Autograft by Dr. Catherine Robertson at UC San Diego
* At least 18 years of age
* Able to Provide Consent in English prior to Surgery

Exclusion Criteria:

* Pregnancy (a urine pregnancy test is standard at UCSD for female patients prior to menopause who are sexually active with the opposite sex within the previous year)
* Inability to communicate with the investigators and hospital staff
* Severe renal, hepatic or cardiac disease
* Chronic high-dose opioid use (defined as daily use for more than 4 weeks prior to surgery of at least the equivalent of 20 mg oxycodone)
* BMI > 45 kg/m2
* Allergy to study medications (lidocaine, bupivacaine)
* Incarceration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Median Post Anesthesia Recovery Unit (PACU) Pain Score | From arrival in PACU until patient has been cleared for PACU discharge
  Median pain score collected in the PACU following surgery on a scale of 1-10 (1 being no pain, 10 being the worst pain the patient has ever experienced)
Total Perioperative Opioid Use (Morphine equivalents) | From time of the start of surgery until time that patient meets PACU discharge criteria
  Intraoperative and Post Operative (in the PACU) opioid use

SECONDARY OUTCOMES:
PACU Length of Stay (days) | From PACU arrival until criteria for PACU discharge are met
  Length of stay from PACU arrival to "ready for discharge" criteria are met
PACU Opioid Use (Morphine equivalents) | From PACU arrival until criteria for PACU discharge are met
  All opioid use in the PACU
Postoperative Day (POD) 1 Opioid Use (Morphine Equivalents) | Time of discharge from PACU until 24 hours after PACU discharge
  All Opioid use in the approximate 24 hours following PACU Discharge
Best, Worst, Average Pain Scores on POD 1 | For the entire length of post operative day 1
  Best, Worst and Average pain scores collected on POD 1 following surgery on a scale of 1-10 (1 being no pain, 10 being the worst pain the patient has ever experienced)

IPD SHARING:
Plan to Share IPD: No